CLINICAL TRIAL: NCT04492501
Title: Role of Investigational Therapies Alone or in Combination to Treat Moderate, Severe and Critical COVID-19
Brief Title: Investigational Treatments for COVID-19 in Tertiary Care Hospital of Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNICEF (Other)
Collaborators: Pak Emirates Military Hospital Rawalpindi (Unknown)
Responsible Party: Principal Investigator, sultan mehmood kamran, Classified Medical specialist, UNICEF
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Sultan Mehmood Kamran 3
Record Dates: First submitted 2020-07-28; First posted 2020-07-30 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Covid19; Cytokine Release Syndrome; Critical Illness; ARDS
Keywords: Therapeutic Plasma exchange; tocilizumab; remdesivir; convalescent plasma; mesenchymal stem cell; COVID-19; investigational treatment
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Critical Illness | interventions — Plasma Exchange; tocilizumab; remdesivir

STUDY DESIGN:
Intervention Model Description: It will be an interventional retrospective case control, single centre based cohort study in Pak Emirates Military Hospital Rawalpindi (PEMH), Pakistan from 1st April to 31st July 2020. This study will be carried out at the Department of Pulmonology and Critical care. PEMH is the largest Covid-19 designated hospital in the country. Data of all hospitalized patients is maintained by PEMH Covid-19 Research and evaluation cell. The study was approved by Institutional Review Board.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Supportive Arm (No Intervention): As per Institutional COVID-19 Management Guidelines all patients of moderate, severe and critical COVID-19 received standard protocol of aspirin, anticoagulation, ulcer prophylaxis, awake Proning (if PaO2 < 80mmHg) and corticosteroids. All patients of Cytokine release storm (CRS) received either Methylprednisolone 1 mg/kg or Dexamethasone 6-12mg/day irrespective of disease severity.
- TPE arm (Experimental): addition to standard care TPE will be performed once daily using COBE Spectra Apheresis machine version 7 (Manufacturer TERUMO BCT, Lakewood, CO, USA INC) having continuous flow centrifugation. Venous access will be achieved using an ultrasound guided double lumen catheter (Arrow - 12 FR) via femoral vein. Patient's total blood volume will be calculated as per Nadler's formula. Anticoagulant acid dextrose ratio will be 1:10 and flow rate 30-40 ml/minutes (Adjusted as per hemodynamic status). Patients' blood pressure, pulse, oxygen saturation will be monitored throughout procedure. Duration of procedure varied from 2-4 hours and 1-1.5 times total plasma volume will be removed during each procedure. Replacement fluid will be fresh frozen plasma (FFP) and normal saline in 2:1 respectively. All procedures will be performed in intensive care or high dependency unit by Apheresis Department of PEMH. TPE will be continued till recovery.
  Interventions: Procedure: Therapeutic Plasma exchange
- TPE in combination with other investigational treatments (Experimental): During TPE, Replacement fluid will be fresh frozen plasma (FFP) and normal saline in 2:1 respectively plus 200-400 ml of convalescent plasma. A predefined number of patients will also receive mesenchymal stem cell therapy and/or Remdesivir
  Interventions: Procedure: Therapeutic Plasma exchange; Biological: Convalescent Plasma; Drug: Tocilizumab; Drug: Remdesivir; Biological: Mesenchymal stem cell therapy
- Either alone or combination of MSC, Remdesivir and Tocilizumab (Experimental): A predefined number of patients will receive either alone Tocilizumab, Remdesivir and Mesenchymal stem cell therapy or their combination
  Interventions: Procedure: Therapeutic Plasma exchange; Biological: Convalescent Plasma; Drug: Tocilizumab; Drug: Remdesivir; Biological: Mesenchymal stem cell therapy

INTERVENTIONS:
Procedure: Therapeutic Plasma exchange — 1-1.5 plasma volume exchange, 2/3rd plasma should be replacing with FFP to avoid coagulopathy, adequate dieresis to prevent volume overload, 1-5 sessions in total, 1 session daily
  Arms: Either alone or combination of MSC, Remdesivir and Tocilizumab; TPE arm; TPE in combination with other investigational treatments
Biological: Convalescent Plasma — Convalescent plasma as part of replacement therapy (200-400ml) if reported within 14 days of illness. An IgG titer of > 1.320 will be considered suitable for use. It will be Collected from person previously infected with Covid-19 and meet following criteria;
  1. After 28 day of illness till 3 months
  2. Symptom free 2 weeks prior to donation
  3. Negative two consecutive PCRs any time between initial positivity and before donation
  4. Anti SARS-CoV2 IgG positive, IgM negative
  5. Fulfills healthy donor criteria as per WHO/AABB guidelines
  6. Volume of plasma to be collected: 900-1200 ml through Apheresis OR plasma separated from phlebotomy donation
  Arms: Either alone or combination of MSC, Remdesivir and Tocilizumab; TPE in combination with other investigational treatments
Drug: Tocilizumab — A predefined number of patients having evidence of cytokine release storm with normal procalcitonin level for three consecutive days, a normal blood culture and IL-6 level > 3 times ULN will be given 1-2 doses of Tocilizumab (80mg IV) . Following contraindications to Tocilizumab will be considered (Allergy to any monoclonal Ab, ANC < 1000, Platelets < 50, ALT or AST > 5 times ULN, Pregnancy and breast feeding, Post TB lung). Some patients will receive it alone in addition to standard treatment whereas in few patients where indicated it will be given in combination with MSC or Remdesivir or both
  Arms: Either alone or combination of MSC, Remdesivir and Tocilizumab; TPE in combination with other investigational treatments
Drug: Remdesivir — It will be given to selected patients who have evidence of hypoxemia and presented with in 14 days of illness. For adults requiring invasive mechanical ventilation the dosage of remdesivir is a single loading dose of 200 mg sta on Day 1 followed by once daily maintenance doses of 100 mg IV for 9 days (days 2 through 10). For adults not requiring invasive mechanical ventilation 5 standard doses will be used. However, patients with known hypersensitivity to Remdesivir, multi organ failure, ALT > 5 times ULN and GFR < 30ml/minute will not be given Remdesivir. In some patients, where indicated other novel treatments including MSC therapy, Tocilizumab and therapeutic plasma exchange will be given.
  Arms: Either alone or combination of MSC, Remdesivir and Tocilizumab; TPE in combination with other investigational treatments
Biological: Mesenchymal stem cell therapy — Single Dose of 2 x 106 cells/kg will be administered either alone or in combination with other novel therapies. At Armed Forces Bone Marrow Transplant Centre (AFBMTC), MSCs will be isolated from bone marrow harvested cells. About 50ml bone marrow will be collected from iliac crest using aseptic technique in syringes primed with anticoagulant. The collected sample will be diluted with Phosphate Buffer Saline (PBS) and MSCs will be separated using density gradient centrifugation. After resuspension the cells will be seeded at a fixed concentration of 100,000 cells/cm2 in specially designed flasks and incubated at 37Oc in 5% CO2. Medium will be changed after every third day till harvesting of MSCs from the flasks. Once confluent (approximately day 20) the cells will be harvested with sterile techniques using Trypsin- EDTA solution.
  Other Names: MSC
  Arms: Either alone or combination of MSC, Remdesivir and Tocilizumab; TPE in combination with other investigational treatments

SUMMARY:
Beyond supportive care, there are currently no proven treatment options for coronavirus disease (COVID-19) and related pneumonia, caused by Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2).Investigators have seen recently from experience in Western countries with best health care systems that pandemics cannot be managed in hospitals. Investigators have seen ICUs crowded to capacity, healthcare workers being exposed and going to quarantine or dying after exposure to large doses of viral inoculums. Investigators recommend that institutions should register for Clinical trials and consider emergency use of TPE. In Pandemics, time is of essence to avoid mortality by intervening early with available evidence, preferably as part of clinical trial.Since the outbreak of corona virus disease (COVID-19), main treatment modalities have been antivirals, interferons, glucocorticoids, anti-coagulants and supportive treatment in addition to traditional Chinese medicine. There are also clinical trials exploring hydroxyquinoline / chloroquine sulphate, azithromycin, immunoglobulins, Vitamin-C, washed microbiota, nebulized interferon, teicoplanin as well as Mesenchymal stem cells. However, most of these trials were small and remain in the experimental phase with currently no effective / speciﬁc antiviral with robust scientific evidence as regards the mortality reduction in COVID-19.In an attempt to treat COVID-19, investigator will use different investigational treatment either alone or in combination to see mortality and morbidity benefit on the basis of limitted evidence available so far. These investigational modalities include Therapeutic plasma exchange (TPE), Convalescent Plasma (CP), Remdesivir, Tocilizumab and Mesenchymal stem cell (MSC) therapy in addition to standard supportive treatment.

DETAILED DESCRIPTION:
Long title: Role of different investigational treatments alone or in combination to treat moderate, severe and critical COVID-19 in addition to standard treatment; An Open label, Phase 2 Study Clinical Phase: multi arm, Phase 2 Open Label Conducted by: Department of Pulmonology and Critical Care; Pak Emirates Military Hospital. Sample Size: 600 Study Population: Hospitalized COVID-19 patients aged ≥18 years to 80 years of with Moderate- severe-critical disease Study Duration: 1st April, 2020 to 31st July 2020 Study Design: This open label phase 2 trial will assess the efficacy and safety of following treatment options 1. Standard treatment including steroids 2. Therapeutic plasma exchange in addition to standard treatment 3. Therapeutic Plasma exchange in combination with Convalescent Plasma in addition to standard treatment 4. Tocilizumab in addition to standard treatment 5. Remdesivir alone or in combination with Therapeutic plasma exchange in addition to standard treatment 6. Mesenchymal stem cell therapy in combination with other investigational treatments in addition to standard treatment Operational Definitions

1. Moderate disease:

   COVID-19 positive case with lung infiltrates < 50% of total lung fields on Chest X-ray / peripheral ground glass opacities (GGOs) on High Resolution Computerized Tomography (HRCT)chest but no evidence of hypoxemia.
2. Severe disease:

   COVID-19 pneumonia with evidence of hypoxemia (RR > 30/minute or PaO2 on ABGs < 80mmHg or PaO2/FiO2 (PF ratio) < 300 or lung infiltrates > 50% of the lung field).
3. Critical illness:

   COVID-19 pneumonia with evidence of either respiratory failure (PaO2 < 60mmHg) or multiorgan dysfunction syndrome (MODS) measured by Sequential Organ Failure assessment (SOFA score) > 10 or septic shock (Systolic BP less than 90 or less than 40mm Hg of baseline in hypertensive or Urine output < 0.5 ml/kg/hour).Age, sex, comorbidities, date of symptoms, source of infection, type of admission SOFA score, Clinical status, vital signs including temperature, respiratory rate, oxygen saturation, oxygen requirement, Complete Blood counts (CBC) with neutrophil counts, lymphocytes count, C-reactive Proteins (CRP), chest imaging (CT or X-ray), location and status in hospital
4. Cytokine release storm (CRS):

Diagnostic criteria of Cytokine release syndrome (CRS) CRS is defined as fever of equal to or more than 100 F persisting > 48 hours in absence of documented bacterial infection and ANY of the following in the presence of moderate, severe or critical disease

1. Ferritin >1000 mcg/L and rising in last 24 hours
2. Ferritin >2000 mcg/L in patient requiring high flow oxygen or ventilation
3. Lymphopenia < 800 cells/ul or lymphocyte percentage <20% and two of the following

   1. Ferritin >700 mcg/mL and rising in the last 24 hours
   2. LDH > 300 IU (reference 140-250 IU/L) and rising in the last 24 hours
   3. D-Dimer >1000ng/mL (or >1mcg/ml) and rising in the last 24 hours
   4. CRP >70 mg/L (or >10 hsCRP) and rising in the last 24 hours, in absence of bacterial infection
   5. If any 3 of above presents on admission no need to document rise

5. Standard treatment: As per Institutional COVID-19 Management Guidelines all patients of moderate, severe and critical COVID-19 received standard protocol of aspirin, anticoagulation, ulcer prophylaxis, awake Proning (if PaO2 < 80mmHg) and corticosteroids. All patients of CRS received Methylprednisolone 1 mg/kg irrespective of disease severity. 6. Therapeutic Plasma exchange (TPE) Therapeutic plasma exchange: 1-1.5 plasma exchange daily (1-5 sessions) with replacement fluid Fresh frozen Plasma (FFP) (whole volume) to 70 willing patients of moderate, severe and critical disease with evidence of CRS after explaining the investigational role of this therapy. TPE will be given in addition to standard treatment to 70 patients randomly. TPE related complications to be documented 7. Recovery Recovery to be defined by de-escalation of patients condition from severe to moderate, or from moderate to mild, plus at least 2 of the following; serum Ferritin < 1000 ug/ml (and decreasing trend on two consecutive days), serum LDH normalization, C-reactive protein > 50% fold reduction (and decreasing trend in on two consecutive days),), ALC > 1000 and PT/APTT normalization.

ELIGIBILITY:
Inclusion Criteria:

* PCR positive confirmed COVID-19
* Admitted in hospital
* willing patients to participate in trial
* Day of illness less than 14 days
* no contraindications to invasive procedure or novel therapies

Exclusion Criteria:

* co morbidities with life expectancy less than 6 months
* Multi organ failure
* Septic shock before initiation of treatment
* Congestive cardiac failure (EF<20%) (4)
* Those receiving immunotherapy, Anti-thymocyte globulin or hematopoietic stem cell transplant in recent past
* Patients of hematological or solid organ malignancies

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-07-20 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
survival | 28 days
  death or recovery

SECONDARY OUTCOMES:
duration of hospitalization | 28 days
  duration in days
Time to resolution of cytokine release storm | 28 days
  duration in days to normalize symptoms and laboratory parameters
Time of viral clearance | 45 days
  Time in days to turn PCR negative
Complications | 90 days
  incidence of Post Covid lung fibrosis

CONTACTS AND LOCATIONS:
Overall Officials: Sumaira Irum, MIT, Study Director — UNICEF
Locations (1):
- Pak Emirates Military Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
data can be shared on demand in SPSS sheet
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months from completion of study
Access Criteria: email

REFERENCES:
- [Background] Knaup H, Stahl K, Schmidt BMW, Idowu TO, Busch M, Wiesner O, Welte T, Haller H, Kielstein JT, Hoeper MM, David S. Early therapeutic plasma exchange in septic shock: a prospective open-label nonrandomized pilot study focusing on safety, hemodynamics, vascular barrier function, and biologic markers. Crit Care. 2018 Oct 30;22(1):285. doi: 10.1186/s13054-018-2220-9. PMID 30373638
- [Background] Keith P, Day M, Perkins L, Moyer L, Hewitt K, Wells A. A novel treatment approach to the novel coronavirus: an argument for the use of therapeutic plasma exchange for fulminant COVID-19. Crit Care. 2020 Apr 2;24(1):128. doi: 10.1186/s13054-020-2836-4. No abstract available. PMID 32241301
- [Background] Shi H, Zhou C, He P, Huang S, Duan Y, Wang X, Lin K, Zhou C, Zhang X, Zha Y. Successful treatment with plasma exchange followed by intravenous immunoglobulin in a critically ill patient with COVID-19. Int J Antimicrob Agents. 2020 Aug;56(2):105974. doi: 10.1016/j.ijantimicag.2020.105974. Epub 2020 Apr 13. PMID 32298745
- [Background] Chen L, Xiong J, Bao L, Shi Y. Convalescent plasma as a potential therapy for COVID-19. Lancet Infect Dis. 2020 Apr;20(4):398-400. doi: 10.1016/S1473-3099(20)30141-9. Epub 2020 Feb 27. No abstract available. PMID 32113510
- [Background] Xu X, Han M, Li T, Sun W, Wang D, Fu B, Zhou Y, Zheng X, Yang Y, Li X, Zhang X, Pan A, Wei H. Effective treatment of severe COVID-19 patients with tocilizumab. Proc Natl Acad Sci U S A. 2020 May 19;117(20):10970-10975. doi: 10.1073/pnas.2005615117. Epub 2020 Apr 29. PMID 32350134
- [Background] Beigel JH, Tomashek KM, Dodd LE, Mehta AK, Zingman BS, Kalil AC, Hohmann E, Chu HY, Luetkemeyer A, Kline S, Lopez de Castilla D, Finberg RW, Dierberg K, Tapson V, Hsieh L, Patterson TF, Paredes R, Sweeney DA, Short WR, Touloumi G, Lye DC, Ohmagari N, Oh MD, Ruiz-Palacios GM, Benfield T, Fatkenheuer G, Kortepeter MG, Atmar RL, Creech CB, Lundgren J, Babiker AG, Pett S, Neaton JD, Burgess TH, Bonnett T, Green M, Makowski M, Osinusi A, Nayak S, Lane HC; ACTT-1 Study Group Members. Remdesivir for the Treatment of Covid-19 - Final Report. N Engl J Med. 2020 Nov 5;383(19):1813-1826. doi: 10.1056/NEJMoa2007764. Epub 2020 Oct 8. PMID 32445440
- [Background] Leng Z, Zhu R, Hou W, Feng Y, Yang Y, Han Q, Shan G, Meng F, Du D, Wang S, Fan J, Wang W, Deng L, Shi H, Li H, Hu Z, Zhang F, Gao J, Liu H, Li X, Zhao Y, Yin K, He X, Gao Z, Wang Y, Yang B, Jin R, Stambler I, Lim LW, Su H, Moskalev A, Cano A, Chakrabarti S, Min KJ, Ellison-Hughes G, Caruso C, Jin K, Zhao RC. Transplantation of ACE2- Mesenchymal Stem Cells Improves the Outcome of Patients with COVID-19 Pneumonia. Aging Dis. 2020 Mar 9;11(2):216-228. doi: 10.14336/AD.2020.0228. eCollection 2020 Apr. PMID 32257537